CLINICAL TRIAL: NCT04399642
Title: Intra-articular Vancomycin Powder in Knee and Hip Arthroplasty: a Prospective, Randomized Clinical Survey
Brief Title: Intra-articular Vancomycin Powder in Knee and Hip Arthroplasty
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other)
Responsible Party: Principal Investigator, Benoit Benoit, Orthopaedic surgeon, principal investigator, Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Single-Dose
Record Dates: First submitted 2020-05-15; First posted 2020-05-22 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Infection
Keywords: vancomycine; hip arthroplasty; knee arthroplasty; hip revision arthroplasty; knee revision arthroplasty
MeSH Terms: conditions — Infections | interventions — Arthroplasty; Arthroplasty, Replacement, Knee; Arthroplasty, Replacement, Hip

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Because of the nature of the intervention, it is impossible for the surgeon to be blinded. However, postoperative infection will be diagnosed by an independent co-worker, not involved in the surgery. Patients will be blind as they will not be aware if they had intra-articular vancomycin powder or not
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard (Active Comparator): Patients receiving single dose of IV cefazolin (2 grams if < 120kg; 3 grams if >120kg) 10-60 minutes before incision
  Interventions: Procedure: Arthroplasty
- Vanco (Experimental): Patients receiving a single dose of IV cefazolin (2 grams if < 120kg; 3 grams if >120kg) 10-60 minutes before incision + a single dose of intra-articular vancomycin powder (1 gram) before articulation (hip or knee) closure
  Interventions: Procedure: Arthroplasty

INTERVENTIONS:
Procedure: Arthroplasty — All patients include in the study will undergo a lowerlimb arthroplasty, primary or revision
  Other Names: Knee arthroplasty; Hip arthroplasty; Knee aseptic revision arthroplasty; Hip arthroplaty revision

SUMMARY:
The purpose of this study is to compare infection rates when patients, elected for primary or aseptic revision THA / TKA, have a single intravenous antibiotic dose versus one single intravenous antibiotic dose in combination with intra-articular antibiotics. This is a prospective, randomized clinical survey on selected outcome measurements on 1834 subjects who will be recruited in a period of about 2 years.

DETAILED DESCRIPTION:
Group A: patients receiving single dose of IV cefazolin 10-60 minutes before incision.

Group B: patients receiving a single dose of IV cefazolin 10-60 minutes before incision + a single dose of intra-articular vancomycin powder before articulation (hip or knee) closure.

ELIGIBILITY:
Inclusion Criteria:

* Standard criteria for the implantation of primary total hip or knee replacement
* Revision of an aseptic THA or TKA.
* Adults >18 years of age
* Diagnosis of Osteoarthrosis (OA), Osteonecrosis (ON), Arthritis; or aseptic loosening of THA/TKA.
* Subject is willing to consent to participate in the study
* Subject is available for follow-up through at least 2 years
* Subject has met acceptable preoperative medical clearance and is free of or treated for medical conditions that would pose excessive operative risk.
* Subject who are fluent in English and / or French and able to understand their role in the study

Exclusion Criteria:

* Active, local infection or systemic infection.
* Participation in any other pharmaceutical, biologic or medical device clinical investigation
* Subjects with known allergy to vancomycin
* Subjects unable to consent
* Patient with skin pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1832 (Estimated)
Dates: Start 2019-07-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Acute Infection rate | 3 months
  Infection rate after after lowerlimb arthroplasty depending on the antibiotic molecule that was given

SECONDARY OUTCOMES:
Long-term infection rate | 2 years
  Infection rate after after lowerlimb arthroplasty depending on the antibiotic molecule that was given
Risk factor | 2 years
  Infection rate in patients with risk factors depending on the antibiotic molecule that was given
Primary vs revision | 2 years
  Infection rate in primary versus revisions surgery depending on the antibiotic molecule that was given
Surgery time | 2 years
  Infection rate according to surgery time depending on the antibiotic molecule that was given

OTHER OUTCOMES:
The Western Ontario and McMaster Universities Arthritis Index (WOMAC) | baseline, 1 year
  Scale from 0 to 97. 97 indicate worse pain, stiffness, and functional limitations
EQ-5D-5L | baseline, 1 year
  The descriptive system section of the EQ-5D questionnaire produces a 5-digit health state profile that represents the level of reported problems on each of the five dimensions of health

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Benoit, MD, Principal Investigator — CIUSSS du Nord de l'Île de Montreal
Locations (1):
- Hopital Sacré-Coeur de Montreal, Montreal, Quebec, Canada